CLINICAL TRIAL: NCT07328568
Title: The Effect of Low Volume Sprint Interval Training on Cardiorespiratory Fitness--a Randomized Controlled Trial
Brief Title: Effect of Low Volume Sprint Interval Training on Cardiorespiratory Fitness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, San Marcos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R15AG093525 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Inactivity, Physical; Overweight (BMI > 25); Healthy Participants
Keywords: high intensity interval training; maximal oxygen uptake; fat metabolism; affective valence; body composition; exercise adherence
MeSH Terms: conditions — Sedentary Behavior; Overweight | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial.
Masking Description: Investigators are masked to participant randomization which is performed by an individual who has no interaction with participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will perform long term REHIT.
  Interventions: Other: High intensity interval training
- Non exercising control group (Placebo Comparator): This group will not complete REHIT, and will be given the option to complete the training once post testing is performed.
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: High intensity interval training — Participants will complete 24 sessions of REHIT and their responses will be compared to a non exercising control group.

SUMMARY:
Low levels of physical activity (PA) are related to poor health and greater risk of premature death in adults. Lack of time is cited as a primary barrier to partaking in PA. In the last 20 years, a lot of attention has been directed towards the efficacy of high intensity interval training (HIIT), which consists of brief, intense bursts of PA separated by recovery. One primary benefit of HIIT is a sizable increase in cardiorespiratory fitness (CRF), which enables adults to exercise better and reduce health risks due to the strong link between health status and CRF.

Completion of cardiovascular exercise is typically recommended for all adults to increase CRF, yet it takes a lot of time and may be perceived as boring. Alternatively, HIIT requires less time and tends to cause greater feelings of enjoyment in many adults. Hundreds of studies report an increase in CRF in response to HIIT in various groups of adults ranging from athletes and those with obesity, diabetes, cancer, stroke, and even spinal cord injury, which emphasizes the potency of this vigorous form of PA. Yet, many studies are weakened by a small sample size which questions the feasibility of these findings.

This randomized controlled trial will test the efficacy and feasibility of a very small amount of HIIT, referred to as reduced exertion high intensity interval training (REHIT), in inactive adults. In the proposed study, REHIT will consist of 2 days per week of 1 to two 10 - 20 second sprints on a stationary bike. The proposed sample will include 60 adults who complete 18 sessions of REHIT over a 9 week period, and their responses will be compared to a non exercising control group. During the study, changes in CRF, fuel metabolism, and psychological responses will be monitored, with the latter outcome shedding light on the overall feasibility of HIIT in inactive adults.

Overall, this novel study has profound public health applications as it will assess fitness and health related changes to a small dose of PA in the largest sample to date. If substantial changes in CRF are shown, these data have the potential to modify public health guidelines for implementing PA in inactive adults.

DETAILED DESCRIPTION:
Low levels of physical activity (PA) and cardiorespiratory fitness (CRF) are significant issues for societal health. Public health guidelines for adults recommend > 150 min of moderate-intensity continuous training (MICT) or 75 min of vigorous exercise per week, and strength training on > 2 days per week. However, in 2020, 75% of adult Americans did not meet these PA recommendations. Physical inactivity is the fourth leading cause of death worldwide, as it increases the risk of 40 chronic conditions. Low maximal oxygen uptake (V̇O2max; the gold standard index of CRF) is strongly associated with increased risk of future morbidity and all-cause mortality. In fact, many large-scale studies have reported V̇O2max to be a more powerful predictor of risk for future morbidity and all-cause mortality than more traditional risk factors such as smoking, hypertension, obesity, high cholesterol, and insulin resistance. For population-level health, the largest benefits from improved PA and CRF are gained by the least fit individuals, with even small increases in fitness shown to improve health. Despite exercise being the only viable means to improve V̇O2max, it remains underutilized for primary disease prevention. Nevertheless, adults do not engage in PA due to a perceived lack of time. High intensity interval training (HIIT) is a time-efficient form of PA requiring brief intense bursts of activity separated by rest periods. Empirical data show that HIIT elicits similar and in some cases superior benefits versus MICT, often with less time. A special type of HIIT is reduced exertion high intensity interval training (REHIT) requiring only two 20 second sprints within a 10 minute session. A few studies show that REHIT increases CRF and other health-related outcomes, yet these studies have been criticized due to their small sample size, which serves to question the broad application of REHIT in adults. The proposed randomized controlled trial will recruit 60 inactive adults to complete 24 sessions of REHIT and compare resultant changes in CRF, substrate metabolism, and psychological responses to a non-exercising control group. This sample size is threefold higher than used in prior work and provides adequate statistical power to detect meaningful increases in V̇O2max. The proposed study will advance further research in the area of HIIT and if successful, may promote inclusion of REHIT in PA recommendations as a feasible alternative or adjunct to moderate or vigorous-intensity exercise as promoted in current PA recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI < 35 kg/m2
* younger than 65 yr old
* no joint issues

Exclusion Criteria:

* Those adults who are currently active and not weight stable
* Adults with BMI > 35 kg/m2
* Use of medications which may alter study outcomes

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | CRF will be assessed at baseline 48 - 72 hours before the start of training, and at 6 and 12 weeks of training, which represent halfway and end of training. The assessments will be performed at least 24 hours after sessions of exercise training.
  Cardiorespiratory fitness (CRF) is determined by oxygen transport from cardiovascular system to mitochondria and is strongly related to health status and premature mortality. It will be assessed using VO2max testing on a cycle ergometer and expressed in mL/kg/min.

SECONDARY OUTCOMES:
Fat and Carbohydrate Oxidation | Fat and carbohydrate oxidation will be measured at baseline before the start of training and at 6 and 12 weeks of training, representing halfway and end of training, and at baseline and at 12 weeks in the non exercising control group.
  Substrate metabolism represents the breakdown of fat and carbohydrate for energy expenditure and is related to metabolic health. It is measured during submaximal exercise during which time, participants' expired air is collected continuously. In this study, participants will complete 10 min of low intensity exercise before the VO2max test, and gas exchange data will be acquired to estimate the respiratory exchange ratio (RER) which is used to assess the percent contribution of fat and carbohydrate use. Moreover, fat and CHO oxidation will be calculated from standard equations and expressed in g/min.
Cardiac output | CO will be measured at baseline and at 6 and 12 weeks of training, representing halfway and the end of training, and at baseline and at 12 weeks in the non exercising control group.
  Cardiac output (CO in L/min) refers to the amount of blood delivered by the heart each minute and is the product of stroke volume and HR. Its assessment can shed light on the factors explaining the increase in VO2max with exercise training. In this study, it will be measured noninvasively using thoracic impedance cardiography.
Enjoyment of REHIT | This outcome will be assessed during session #2 of each week of training in the exercise training group. So, this outcome will be assessed weekly during all 12 weeks of training.
  The real-world feasibility and efficacy of REHIT has been challenged, as it is thought that this type of vigorous exercise is not enjoyable for adults. One measure related to this is enjoyment, which can be assessed with the 18-item Physical Activity Enjoyment scale. This validated survey is frequently used in similar studies to gauge psychological responses to exercise training. The Physical Activity Enjoyment scale will be completed 5 minutes after sessions of exercise training.
Perceived exertion responses to REHIT | This outcome will be assessed during session #2 of each week of training in the exercise training group. So, this outcome will be assessed weekly during all 12 weeks of training
  The real-world feasibility and efficacy of REHIT has been challenged, as it is thought that this type of vigorous exercise is not enjoyable for adults. One measure related to this is perceived exertion, which can be assessed with the 6 - 20 Borg scale of Rating of Perceived Exertion. This validated survey is frequently used in similar studies to gauge psychological responses to exercise training. This RPE scale will be administered throughout sessions of exercise training, including at baseline, during the warm-up, after sprint 1, midway during recovery, after sprint 2, and then at the end of the exercise session.
Pleasure responses to REHIT | This outcome will be assessed during session #2 of each week of training in the exercise training group. So, this outcome will be assessed weekly during all 12 weeks of training
  The real-world feasibility and efficacy of REHIT has been challenged, as it is thought that this type of vigorous exercise is not pleasing for adults which may cause poor adherence to training. One measure related to this is pleasure:displeasure, which can be assessed with the +5 to -5 Feeling Scale, where +5 = very good, 0 = neutral, and -5 is very bad. This validated survey is frequently used in similar studies to gauge psychological responses to exercise training. This Feeling Scale will be administered throughout sessions of exercise training, including at baseline, during the warm-up, after sprint 1, midway during recovery, after sprint 2, and then at the end of the exercise session.

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Astorino, Ph.D, Principal Investigator — California State University, San Marcos
Locations (1):
- California State University--San Marcos Human Performance Laboratory, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be reported in articles published related to this project.

DOCUMENTS (2):
  • Statistical Analysis Plan: Data analysis (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT07328568/SAP_000.pdf
  • Informed Consent Form: Consent form (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT07328568/ICF_001.pdf